CLINICAL TRIAL: NCT05672979
Title: Prospective triAl of Modified Treat-and-extend Regimens With BroLucizumab in pachychOroid Neovasculopathy
Acronym: PABLO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Min Sagong, Professor, Yeungnam University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YUMC 2022-11-016
Record Dates: First submitted 2022-12-21; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Age-Related Macular Degeneration; Pachychoroid Neovasculopathy
MeSH Terms: conditions — Macular Degeneration | interventions — brolucizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brolucizumab treated (Experimental): Intravitreal brolucizumab 6mg injection.
  Initial treatment consists of a loading dose of three intravitreal injections of brolucizumab at monthly intervals. After 3 loading doses, patients are followed by monthly observation visits until the month 6 and bimonthly afterwards until disease-recurrence interval is determined (It can be monthly as per the investigator's judgement.). Following loading phase, the first treatment interval is determined by patients' disease recurrent interval, 1 month shorter than first recurrence interval (maximum first injection interval is 16 weeks). The injection interval is shortened if there is any fluid change or decreased visual acuity. If the criteria for treatment adjustment were not met and residual fluid was decreased from the previous visit, the injection interval is maintained. And the interval is extended if there was no fluid on OCT. The minimum and maximum injection intervals are 8 and 16 weeks, respectively.
  Interventions: Drug: Brolucizumab Injection [Beovu]

INTERVENTIONS:
Drug: Brolucizumab Injection [Beovu] — brolucizumab 6mg intravitreal injection

SUMMARY:
PNV is a recently described clinical entity; therefore, studies about treatment efficacy and safety are few, with limited follow-up and a small number of participants. Treatment is based on intravitreal anti-VEGF injections, similar to neovascular AMD. According to reported results however, efficacy seems different in fluid reabsorption among anti-VEGF agents. A newly developed anti-VEGF molecule for the treatment of neovascular AMD, brolucizumab, has been shown in clinical studies to have longer durability and improved visual outcomes using a q12-week regimen, thus having the potential to reduce treatment burden and serve as an important therapeutic tool in the management of neovascular AMD. Nevertheless, there have been no reports specifically focusing on the efficacy of brolucizumab in the treatment of PNV. The purpose of this study is to evaluate the efﬁcacy and safety proﬁle of the modified treat-and-extend regimen to 64 weeks by intravitreal brolucizumab injection in eyes with treatment-naive pachychoroid neovasculopathy (PNV) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Male or female patients ≥ 19 years of age at screening
3. Treatment-na¨ıve pachychoroid neovasculopathy (Minimum cutoff value of SFCT 300 μm)
4. Presence of intraretinal fluid (IRF) or subretinal fluid (SRF) that affects the central subfield, as seen by Spectral Domain Optical Coherence Tomography (SD-OCT) (study eye)
5. Best-corrected visual acuity (BCVA) score between 83 and 23 letters, inclusive, using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at both screening and baseline visit (study eye)
6. If both eyes are eligible as per the inclusion and exclusion criteria described below, the eye with the worse visual acuity should be selected for study eye, unless the Investigator deems it more appropriate to select the eye with better visual acuity, based on medical reasons or local ethical requirements.

Exclusion Criteria:

1. Ocular conditions/disorders at screening or baseline which could, in the opinion of the investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require planned medical or surgical intervention during the first 12-month study period, structural damage of the fovea, atrophy or fibrosis at the center of the fovea (study eye)
2. A history of any evidence of type 2 or type 3 neovascularization, polypoidal choroidal vasculopathy (aneurysmal type-1 neovascularization), myopic choroidal neovascularization, or other ocular disorders requiring anti-VEGF treatment.
3. Any active intraocular or periocular infection or active intraocular inflammation, at screening or baseline (study eye)
4. Uncontrolled glaucoma defined as intraocular pressure (IOP) > 25 mmHg on medication, or according to investigator's judgment, at screening or baseline (study eye)
5. Ocular treatments: previous treatment with any anti-vascular endothelial growth factor (VEGF) drugs or investigational drugs, previous use of intraocular or periocular steroids within the 6-month period prior to baseline, history of any macular laser treatment or PDT, ocular surgery except cataract surgery within 3 months prior to baseline will be excluded.
6. Stroke or myocardial infarction during the 6-month period prior to baseline
7. Uncontrolled blood pressure defined as a systolic value ≥160 mmHg or diastolic value ≥100 mmHg at Screening or Baseline. (In case there is an elevated blood pressure measurement, it should be repeated after 20 minutes. If the repeat measurement is elevated, then the participant is not eligible to be enrolled into the study).
8. Systemic anti-VEGF therapy at any time.
9. History of hypersensitivity to any of the study treatment or its excipients or to drugs of similar chemical classes, or clinically relevant sensitivity to fluorescein dye as assessed by the Investigator.
10. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
11. Use of other investigational drugs within 5 half-lives of Baseline, or within 30 days /until the expected pharmacodynamic effect has returned to Baseline, whichever is longer; or longer if required by local regulations (observational clinical studies solely involving over-the-counter vitamins, supplements, or diets are not exclusionary).
12. Physically absence of fellow eye (last eye)
13. Presence of amblyopia, amaurosis or ocular disorders in the fellow eye with BCVA <20/200 at Screening (except when due to conditions whose surgery may improve visual acuity (VA), e.g. cataract).
14. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during the study treatment administration and for one month after stopping the investigational medication. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to Screening). For female participants on the study, the vasectomized male partner should be the sole partner for that participant Use of oral (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in best corrected visual acuity | Week 32
  Mean change from baseline in best corrected visual acuity

SECONDARY OUTCOMES:
Distribution of the last interval | up to Week 32 and Week 64
  Distribution of the last interval with no disease activity
Distribution of the maximal interval | Week 64
  Distribution of the maximal intervals with no disease activity
Time from the last loading injection to the first visit with no disease activity | Week 64
  Time from the last loading injection to the first visit with no disease activity
Proportion of patients with no disease activity | Week 12
  Proportion of patients with no disease activity
Proportion of patients with complete fluid absorption | Week 12, Week 16
  Proportion of patients with complete fluid absorption

IPD SHARING:
Plan to Share IPD: Undecided